CLINICAL TRIAL: NCT06420375
Title: Treatment of Ulcerative Colitis With Novel Therapeutics
Brief Title: Treatment of UC With Novel Therapeutics
Acronym: TURTLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joshua Korzenik, MD-Director, Brigham and Women's Hospital Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025P000585
Record Dates: First submitted 2024-05-06; First posted 2024-05-20 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ulcerative Colitis Mild; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: This is a crossover study in which each participant will receive active medication for a period of time and placebo for a period of time.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blinded study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Comparator: BRS201 Arm (Active Comparator): In Group 1 of the study, subjects will take oral study drug at 1.2g daily, PO (2.4g with 120mg oral butyrate twice daily (240mg daily) for 4 weeks.
  In Group 2 of the study, subjects will take oral study drug at 1.2g twice daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks.
  In Group 3 of the study, subjects will take oral study drug at 1.2g twice daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks. Subjects will also receive a one time 2.5g dose of study drug at initiation.
  In Group 4 of the study, subjects will repeat the previous conditions of the group that proves to be the most effective.
  Interventions: Drug: BRS201
- Placebo Comparator: Placebo Arm (Placebo Comparator): In Group 1 of the study, subjects will take oral placebo at 1.2g daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks.
  In Group 2 of the study, subjects will take oral placebo at 1.2g twice daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks.
  In Group 3 of the study, subjects will take oral placebo at 1.2g twice daily, PO (2.4g daily) with 120mg oral butyrate twice daily (240mg daily) for 4 weeks. Subjects will also receive a one time 100mg dose of cyanocobalamin at initiation.
  In Group 4 of the study, subjects will repeat the previous conditions of the group that proves to be the most effective.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BRS201 — Groups 1, 2, 3, and 4 will all contain 5 subjects each, with each subject receiving active study drug and placebo in a 3:2 randomized order; 3 will receive active treatment for the first for four weeks followed by placebo for four weeks, while the remaining 2 will receive placebo for four weeks followed by active treatment for four weeks.
  Arms: Active Comparator: BRS201 Arm
Drug: Placebo — Groups 1, 2, 3, and 4 will all contain 5 subjects each, with each subject receiving active study drug and placebo in a 3:2 randomized order; 3 will receive active treatment for the first for four weeks followed by placebo for four weeks, while the remaining 2 will receive placebo for four weeks followed by active treatment for four weeks.
  Arms: Placebo Comparator: Placebo Arm

SUMMARY:
This study is a clinical trial being done to investigate the efficacy of drug BRS201 as a treatment in patients with active mild ulcerative colitis. Participation in this study will take 12 weeks long and the study is structured as a crossover study in which participants will take the study drug for 4 weeks and a placebo drug for 4 weeks in a randomized order in the form of an oral medication. Participation may also involve receiving an IV dose of the medication. The study will require participants to attend 7 study visits, all of which will be conducted at a study site. Participation will involve taking an oral medication twice daily, tracking the medication in a log, and getting blood drawn and giving a stool and urine sample for a few lab tests throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give consent
* Patients with a confirmed diagnosis of UC for > 3 months
* History of ≥ 15 cm of colonic involvement as confirmed by colonoscopy
* Disease activity based on calprotectin > 200
* Allowed medications: mesalamine and sulfasalazine
* Patients with primary sclerosing cholangitis are eligible to enroll

Exclusion Criteria:

* History of uncontrolled hypertension with systolic BP > 140 and systolic BP > 90
* Chronic kidney disease as defined by GFR <55mL/min
* Impaired hepatic function (transaminases elevated > 2.5 x ULN) unless due to PSC
* Evidence of C. difficile (Negative test result within 1 month is acceptable)
* Infectious Colitis or drug induced colitis
* Crohn's Disease or Indeterminate colitis
* Decompensated liver disease
* Patients who are pregnant or breastfeeding
* Use of rectal therapies
* Patients who have a confirmed malignancy or cancer within 5 years
* Congenital or acquired immunodeficiencies
* Other comorbidities including: Diabetes mellitus, systemic lupus
* High likelihood of colectomy in the next 2 months
* Participation in a therapeutic clinical trial in the preceding 30 days or simultaneously during this trial
* Patients with a history or risk of cardiovascular conditions, including arrhythmia, long QT syndrome, congestive heart failure, stroke, or coronary artery disease
* Prohibited medications: Vitamin C, prednisone, immune modulators (including but not limited to azathioprine, 6-mercaptopurine, mycophenolate mofetil, tacrolimus, cyclosporine, thalidomide, interleukin-10, interleukin-11, and Omvoh or mirikizumab-mrkz) and biologics within the past six weeks including anti-TNF agents within the past six weeks, vedolizumab within the past six weeks, ustekinumab Risankizumab), a JAKi (tofacitinib or upadacitinib), or Velsipity (etrasimod) within the past 6 weeks. (The aim is to treat people who are having disease activity and just on mesalamine.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of H2S metabolites in plasma | 4 weeks
  The primary endpoint for this study is the capacity of study drug to reduce metabolites of H2S in plasma from baseline (week 0) compared to the end of active treatment (4 weeks)

SECONDARY OUTCOMES:
Simple Clinical Colitis Activity Index (SCCAI) | 12 weeks
  Clinical symptoms assessed by SCCAI which measures patient reported outcomes on a scale of 0 to 19, where a higher score indicates more severe activity and active disease is a score of 5 or more.
Plasma nitrite, nitrate, or nitrosothiol | 8 weeks
  Correlation between changes in plasma nitrite, nitrate or nitrosothiol levels and fecal calprotectin
Normalization of fecal calprotectin lab measurements | 4 weeks
  The primary endpoint for this study is the capacity of study drug to normalize fecal calprotectin levels from baseline (week 0) compared to end of active treatment (4 weeks).
Change in fecal calprotectin lab measurements | 4 weeks
  Change in fecal calprotectin to < ULN at the end of active treatment
Partial Mayo score | 4 weeks
  Change in partial Mayo scores from baseline to end of active treatment. The partial Mayo score measures disease activity on a scale of 0 to 9, where a higher score indicates more severe disease activity and a score of 1 or less indicated remission.
Measurement of sulfur metabolites in urine | 8 weeks
  Analysis of urine for measurement of thiosulfate, thiocyanate, nitrate and nitrite

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States